CLINICAL TRIAL: NCT04109547
Title: China Multi-regional Clinical Trial: Efficacy and Safety of Oral Semaglutide Versus Placebo in Subjects With Type 2 Diabetes Mellitus Treated With Diet and Exercise Only
Brief Title: A Research Study Comparing a New Medicine Oral Semaglutide to Placebo in People With Type 2 Diabetes
Acronym: PIONEER 11
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9924-4338; U1111-1188-1173 (Other: World Health Organization (WHO)); 2018-002590-22 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral semaglutide 3mg (Experimental): Subjects will remain on 3 mg for the entire treatment period (26 weeks)
  Interventions: Drug: Oral semaglutide
- Oral semaglutide 7mg (Experimental): Subjects will receive 3 mg for for the first 4 weeks, 7 mg for the remainder of the treatment period
  Interventions: Drug: Oral semaglutide
- Oral semaglutide 14mg (Experimental): Subjects will receive 3 mg for the first 4 weeks, 7 mg for the next 4 weeks and 14 mg for the remainder of the treatment period
  Interventions: Drug: Oral semaglutide
- Placebo (oral semaglutide) (Placebo Comparator): Subjects will receive placebo tablets for the entire treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral semaglutide — Tablets to be taken once-daily for 26 weeks
  Arms: Oral semaglutide 14mg; Oral semaglutide 3mg; Oral semaglutide 7mg
Drug: Placebo — Tablets to be taken once-daily for 26 weeks
  Arms: Placebo (oral semaglutide)

SUMMARY:
The study compares 2 medicines for type 2 diabetes: oral semaglutide (a new medicine) and placebo (a dummy medicine). Researchers will test semaglutide to see how well it works compared to placebo. The study will also test if semaglutide is safe. Participants will either get semaglutide or placebo - which treatment is decided by chance. Participants will get 1 tablet a day to take with up to half a glass of water. Participants must take the tablet first thing in the morning on an empty stomach. After taking the tablet, participants must not eat or drink anything for at least 30 minutes. After the 30 minutes, participants can have their first meal of the day and take any other medicines they may need. The study will last for about 8 months (36 weeks). Participants will have 9 clinic visits and 2 phone calls with the study doctor. At all 9 of the clinic visits, participants will have blood samples taken. At 5 of the clinic visits, participants must arrive fasting. This means they cannot eat for 8 hours before the visit. It is fine to drink water up to 2 hours before the visit. This is for some of the blood samples that will be taken at the visit. Women cannot take part if pregnant, breastfeeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female, age above or equal to 18 years at the time of signing informed consent.

For Algeria only: Male or female, age above or equal to 19 years at the time of signing the informed consent.

For Taiwan only: Male or female, age above or equal to 20 years at the time of signing the informed consent.

* Diagnosed with type 2 diabetes mellitus
* HbA1c between 7.0 -10.0% (53-86 mmol/mol) (both inclusive).

Exclusion Criteria:

* - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an highly effective contraceptive method.
* Family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC). Family is defined as a first degree relative.
* History or presence of pancreatitis (acute or chronic).
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening.
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV.
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula(CKD-EPI).
* Subjects with alanine aminotransferase (ALT) above 2.5 x upper limit of the normal (ULN).
* Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (66):
- Algeria (2):
  - Bouzareah Diabetic House Algiers Algeria, Algiers
  - UH of Douera, Algiers
- China (48):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Second Affliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - 900th Hospital of Joint Logistics Support Force, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen Universtiy, Guangzhou, Guangdong
  - The 3rd Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - The 2nd Affiliated Hospital of Shantou Uni Medical College, Shantou, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Handan First Hospital, Handan, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The Second People Hospital of Huai'an, Huai'an, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital of Jiaxing, Jiaxing, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - The second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Jining Medical University, Jining, Shandong
  - The Affiliated Hospital of Qingdao Medical College, Qingdao, Shandong
  - Shanghai Pudong New Area People's Hospital, Pudong New District, Shanghai Municipality
  - Rui Jin Hospital,Shanghai Jiao Tong University School of Med, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji university, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hsopital, Tongji University, Shanghai, Shanghai Municipality
  - The Fifth People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Tongren Hospital Shanghai Jiao Tong Univ. School of Medicine, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - First Affiated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Third Xiangya Hospital of Central South University, Changsha
- Hungary (4):
  - Szent Margit Rendelőintézet Nonprofit Kft., Budapest
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Szent Borbála Kórház, Tatabánya
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- Serbia (2):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Centre Nis, Endocrinology, Diabetes and Metabolism, Niš
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linko Branch, Taoyuan
- Ukraine (7):
  - Clinic of Medical Academy, Dnipro, Dnipro
  - CNI "Khmelnytskyi regional hospital" of KRC, Khmelnytskyi
  - Institute of Endocrinology and Metabolism of AMSU, Kyiv
  - City Hospital #1, Mykolaiv
  - CI "1st City Clinical Hospital of Poltava City Council", Poltava
  - CNI "Ternopil University Clinic" of Ternopil Regio. Council, Ternopil
  - Zaporizhia Regional Clinical Endocrinology Dispensary, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Wang W, Bain SC, Bian F, Chen R, Gabery S, Huang S, Jensen TB, Luo B, Yuan G, Ning G; PIONEER 11 investigators. Efficacy and safety of oral semaglutide monotherapy vs placebo in a predominantly Chinese population with type 2 diabetes (PIONEER 11): a double-blind, Phase IIIa, randomised trial. Diabetologia. 2024 Sep;67(9):1783-1799. doi: 10.1007/s00125-024-06142-3. Epub 2024 Jul 10. PMID 38985162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 52 sites in 3 countries and Region China (China mainland and Taiwan) as follows: China mainland (37 sites), Taiwan (3 sites); Hungary (4 sites), Serbia (2 sites) and Ukraine (6 sites).
Pre-assignment Details: Total of 521 participants with type 2 diabetes mellitus treated with diet and exercise only were randomized 1:1:1:1 to receive once-daily blinded treatment for 26 weeks with oral semaglutide 3, 7 or 14 milligrams (mg), or with placebo. The trial included a 4-week run-in period, a treatment period of 26 weeks and a 5-week follow-up period.
Groups:
- Oral Semaglutide 3 mg: Participants received oral semaglutide 3 mg tablets once daily from week 0 to week 26.
- Oral Semaglutide 7 mg: Participants received oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 26: 3 mg from week 0 to week 4 and 7 mg from week 4 to week 26.
- Oral Semaglutide 14 mg: Participants received oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 26: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 26.
- Placebo: Participants received oral semaglutide matching placebo tablets once daily from week 0 to week 26.
Period: Overall Study
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Started | 130 | 130 | 130 | 131
Treated | 130 | 130 | 129 | 131
Full Analysis Set | 130 | 130 | 130 | 131
Safety Analysis Set | 130 | 130 | 129 | 131
Completed | 126 | 126 | 124 | 124
Not Completed | 4 | 4 | 6 | 7
Not completed — Withdrawal by Subject | 3 | 2 | 6 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo | Total
Number analyzed (Participants) | 130 | 130 | 130 | 131 | 521
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (11) | 52 (11) | 53 (10) | 51 (11) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 41 | 47 | 43 | 189
  Male | 72 | 89 | 83 | 88 | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 130 | 130 | 129 | 131 | 520
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Race: Asian | 97 | 97 | 97 | 98 | 389
  Race: White | 33 | 32 | 33 | 33 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline (week 0) in HbA1c at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all randomized participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 117 | 116 | 106
Percentage of HbA1c | -1.1 (0.7) | -1.5 (0.8) | -1.6 (1.0) | -0.2 (0.9)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Placebo; Test type: Superiority; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.5, 95% CI 2-sided [-1.8 to -1.3]
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; Test type: Superiority; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.4, 95% CI 2-sided [-1.6 to -1.2]
Statistical Analysis 3: Comparison: Oral Semaglutide 3 mg vs Placebo; Test type: Superiority; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.0, 95% CI 2-sided [-1.2 to -0.8]

2. Secondary Outcome: Change From Baseline in Body Weight (Kilograms [kg])
Description: Change from baseline (week 0) in body weight at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 116 | 106
Kg | -1.1 (3.3) | -2.2 (3.4) | -3.1 (3.7) | -1.1 (2.7)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 118 | 116 | 104
milligrams per deciliter (mg/dL) | -19.07 (32.44) | -32.28 (27.95) | -32.50 (24.91) | 0.00 (27.49)

4. Secondary Outcome: Change From Baseline in Fasting 7-point Self-measured Plasma Glucose (SMPG) Profile: Mean 7-point Profile
Description: Change from baseline (week 0) in mean 7-point SMPG profile at week 26 is presented. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 110 | 117 | 115 | 104
mg/dL | -29.4 (29.3) | -43.0 (36.1) | -44.5 (36.9) | -10.3 (37.5)

5. Secondary Outcome: Change From Baseline in Fasting 7-point Self-measured Plasma Glucose Profile: Mean Postprandial Increment (Over All Meals)
Description: Change from baseline (week 0) in fasting 7-point SMPG: Mean postprandial increment (over all meals) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 112 | 117 | 115 | 104
mg/dL | -14.5 (34.2) | -20.0 (39.9) | -27.9 (40.6) | -6.7 (35.6)

6. Secondary Outcome: Change From Baseline in Body Weight (Percentage [%])
Description: Change from baseline (week 0) in body weight (measured in kg) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 116 | 106
Percentage change | -1 (4) | -3 (4) | -4 (5) | -1 (3)

7. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from baseline (week 0) in BMI at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 116 | 106
kilograms per square meter (kg/m^2) | -0.4 (1.2) | -0.8 (1.2) | -1.1 (1.3) | -0.4 (0.9)

8. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Change from baseline (week 0) in waist circumference at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimetres (cm)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 116 | 105
centimetres (cm) | -2.1 (4.5) | -2.2 (4.8) | -2.8 (4.4) | -1.4 (3.3)

9. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Total Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in total cholesterol (measured in mg/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 114 | 104
Ratio of total cholesterol | 0.99 (14.75) | 0.98 (16.62) | 0.94 (19.92) | 1.00 (14.45)

10. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Low-density Lipoprotein (LDL) Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in LDL cholesterol (measured in mg/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 114 | 102
Ratio of LDL cholesterol | 1.00 (29.65) | 1.00 (28.35) | 0.94 (31.12) | 1.00 (25.32)

11. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: High-density Lipoprotein (HDL) Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in HDL cholesterol (measured in mg/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 114 | 102
Ratio of HDL cholesterol | 1.03 (15.78) | 1.02 (15.41) | 1.02 (17.72) | 1.04 (14.61)

12. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Triglycerides (Ratio to Baseline)
Description: Change from baseline (week 0) in triglycerides (measured in mg/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 119 | 114 | 102
Ratio of triglycerides | 0.96 (45.32) | 0.90 (45.56) | 0.87 (51.82) | 0.93 (49.08)

13. Secondary Outcome: Change From Baseline in Short Form-36 Version 2 (SF-36v2) (Acute Version) Health Survey
Description: SF-36 v2.0 is a 36-item, patient-reported survey of patient health. SF-36 measures the participant's overall Health Related Quality of Life on 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) and two component summary scores (physical component summary and mental component summary). Range of score for domains and component summary scores : 1-100 (Higher scores indicated a better health state). Change form baseline in each domain, physical component summary score and mental component summary score at week 26 is presented. A positive change score indicates an improvement since baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a score
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 115 | 106
Units on a score
  Physical functioning | 0.25 (4.83) | 0.97 (5.16) | 0.34 (4.24) | 0.87 (4.98)
  Role physical | 0.34 (5.70) | 0.43 (5.83) | -0.00 (5.02) | 0.33 (7.50)
  Bodily pain | 0.11 (8.72) | -0.86 (8.19) | -0.34 (6.56) | 0.49 (8.40)
  General health | 2.01 (7.14) | 2.51 (7.52) | 1.32 (8.61) | 1.17 (5.91)
  Vitality | 1.23 (7.62) | -0.23 (6.96) | 0.54 (8.02) | 0.49 (6.35)
  Social functioning | 0.22 (6.26) | 0.25 (7.22) | -0.60 (6.18) | 0.98 (7.04)
  Role emotional | 0.46 (6.94) | 0.58 (8.34) | 0.33 (7.03) | -0.04 (9.03)
  Mental health | 0.22 (7.59) | -0.38 (7.96) | -0.30 (7.78) | 0.05 (6.99)
  Physical component score | 0.66 (5.21) | 0.88 (4.98) | 0.39 (4.60) | 0.94 (4.71)
  Mental component score | 0.51 (6.86) | -0.15 (7.65) | -0.10 (6.44) | 0.08 (6.88)

14. Secondary Outcome: Number of Participants Who Achieved HbA1c Less Than (<) 7.0 % (53 Millimoles Per Mole [mmol/Mol]) (American Diabetes Association (ADA) Target) (Yes/no)
Description: Number of participants who achieved HbA1c < 7.0 % (53 mmol/mol) (ADA target) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 117 | 116 | 106
Participants
  Yes | 75 | 100 | 92 | 27
  No | 39 | 17 | 24 | 79

15. Secondary Outcome: Number of Participants Who Achieved HbA1c Less Than or Equal to (<=) 6.5 Percent (48 mmol/Mol) (American Association of Clinical Endocrinologists (AACE) Target) (Yes/no)
Description: Number of participants who achieved HbA1c <= 6.5 percent (48 mmol/mol) (AACE target) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 117 | 116 | 106
Participants
  Yes | 53 | 76 | 76 | 12
  No | 61 | 41 | 40 | 94

16. Secondary Outcome: Number of Participants Who Achieved HbA1c Reduction Greater Than or Equal to (>=) 1 Percent (10.9 mmol/Mol) (Yes/no)
Description: Number of participants who achieved HbA1c reduction >= 1 percent (10.9 mmol/mol) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 117 | 116 | 106
Participants
  Yes | 67 | 89 | 87 | 19
  No | 47 | 28 | 29 | 87

17. Secondary Outcome: Number of Participants Who Achieved Body Weight Loss >= 3 Percent (Yes/no)
Description: Number of participants who achieved body weight loss >= 3 percent (yes/no) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 117 | 116 | 106
Participants
  Yes | 33 | 49 | 62 | 28
  No | 81 | 68 | 54 | 78

18. Secondary Outcome: Number of Participants Who Achieved Body Weight Loss >= 5 Percent (Yes/no)
Description: Number of participants who achieved body weight loss >= 5 percent (yes/no) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 116 | 106
Participants
  Yes | 17 | 29 | 43 | 11
  No | 98 | 90 | 73 | 95

19. Secondary Outcome: Number of Participants Who Achieved Body Weight Loss >= 10 Percent (Yes/no)
Description: Number of participants who achieved body weight loss >= 10 percent (yes/no) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 115 | 119 | 116 | 106
Participants
  Yes | 5 | 7 | 12 | 0
  No | 110 | 112 | 104 | 106

20. Secondary Outcome: Number of Participants Who Achieved HbA1c < 7.0 Percent (53 mmol/Mol) Without Hypoglycaemia (Treatment-emergent Severe or Blood Glucose [BG] Confirmed Symptomatic Hypoglycaemic Episodes) and no Body Weight Gain (Yes/no)
Description: Number of participants who achieved HbA1c < 7.0 percent (53 mmol/mol) without hypoglycaemia (treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes) and no body weight gain (yes/no) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 117 | 116 | 106
Participants
  Yes | 54 | 80 | 84 | 19
  No | 60 | 37 | 32 | 87

21. Secondary Outcome: Number of Participants Who Achieved HbA1c Reduction >= 1% (10.9 mmol/Mol) and Body Weight Loss >= 3 Percent (Yes/no)
Description: Number of participants who achieved HbA1c reduction >= 1% (10.9 mmol/mol) and body weight loss >= 3% (yes/no) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 114 | 117 | 116 | 106
Participants
  Yes | 26 | 43 | 53 | 10
  No | 88 | 74 | 63 | 96

22. Secondary Outcome: Time From First Dose to Initiation of Rescue Medication
Description: Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after randomization and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomization and before last day on trial product. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline (Week 0) to Week 26
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 6 | 3 | 0 | 15
Days | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days are reported as Not available (NA). | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days are reported as NA. |  | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days are reported as NA.

23. Secondary Outcome: Semaglutide Plasma Concentrations
Description: Semaglutide plasma concentrations at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: Week 26: post dose any time
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 86 | 88 | 79
nanomoles per liter (nmol/L) | 4.36 (103.74) | 11.22 (106.34) | 17.71 (232.82)

24. Secondary Outcome: Change From Baseline in Haematology - Haematocrit (Ratio to Baseline)
Description: Change from baseline (week 0) in haematocrit (measured in %) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: Safety analysis set included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haematocrit
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 120 | 117 | 116 | 118
Ratio of haematocrit | 1.00 (7.14) | 1.00 (8.10) | 1.00 (6.15) | 1.00 (14.42)

25. Secondary Outcome: Change From Baseline in Haematology - Haemoglobin (Ratio to Baseline)
Description: Change from baseline (week 0) in haemoglobin (measured in millimoles per liter [mmol/L]) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haemoglobin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 120 | 117 | 116 | 118
Ratio of haemoglobin | 1.01 (6.00) | 1.00 (6.82) | 1.00 (6.17) | 1.00 (7.50)

26. Secondary Outcome: Change From Baseline in Haematology - Leucocytes (Ratio to Baseline)
Description: Change from baseline (week 0) in leucocytes (measured in 10^9 per liter [10^9/L]) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of leucocytes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 120 | 117 | 116 | 118
Ratio of leucocytes | 1.03 (18.79) | 1.01 (22.23) | 1.04 (22.60) | 1.03 (20.80)

27. Secondary Outcome: Change From Baseline in Haematology - Thrombocytes (Ratio to Baseline)
Description: Change from baseline (week 0) in thrombocytes (measured in 10^9/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of thrombocytes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 118 | 115 | 114 | 118
Ratio of thrombocytes | 1.03 (23.24) | 1.01 (17.69) | 1.04 (17.55) | 1.02 (19.98)

28. Secondary Outcome: Change From Baseline in Haematology - Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils
Description: Change from baseline (week 0) in basophils, eosinophils, lymphocytes, monocytes and neutrophils at week 26 is presented. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: 10^9 cells per liters (10^9 cells/L)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 119 | 117 | 116 | 118
10^9 cells per liters (10^9 cells/L)
  Basophils | 0.00 (0.06) | -0.01 (0.06) | -0.01 (0.06) | -0.01 (0.07)
  Eosinophils | 0.01 (0.10) | 0.02 (0.10) | 0.02 (0.12) | 0.01 (0.08)
  Lymphocytes | 0.05 (0.43) | -0.03 (0.49) | -0.09 (0.49) | 0.02 (0.46)
  Monocytes | 0.01 (0.12) | -0.00 (0.16) | 0.01 (0.16) | 0.01 (0.15)
  Neutrophils | 0.18 (0.98) | 0.06 (1.44) | 0.28 (1.19) | 0.21 (1.14)

29. Secondary Outcome: Change From Baseline in Biochemistry - Urea (Ratio to Baseline)
Description: Change from baseline (week 0) in urea (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of urea
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 119
Ratio of urea | 1.02 (21.23) | 1.00 (24.90) | 1.02 (23.12) | 1.07 (23.97)

30. Secondary Outcome: Change From Baseline in Biochemistry - Creatinine (Ratio to Baseline)
Description: Change from baseline (week 0) in creatinine (measured in mg/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatinine
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 116 | 119
Ratio of creatinine | 1.03 (10.39) | 1.02 (13.25) | 1.03 (11.50) | 0.99 (11.49)

31. Secondary Outcome: Change From Baseline in Biochemistry - Alanine Aminotransferase (Ratio to Baseline)
Description: Change from baseline (week 0) in alanine aminotransferase (measured in units per liter [U/L]) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of alanine aminotransferase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 116 | 118
Ratio of alanine aminotransferase | 0.88 (44.27) | 0.89 (45.23) | 0.85 (47.44) | 0.88 (42.72)

32. Secondary Outcome: Change From Baseline in Biochemistry - Aspartate Aminotransferase (Ratio to Baseline)
Description: Change from baseline (week 0) in aspartate aminotransferase (measured in U/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of aspartate aminotransferase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 120 | 120 | 111 | 116
Ratio of aspartate aminotransferase | 0.91 (30.50) | 0.91 (34.42) | 0.90 (35.09) | 0.89 (38.14)

33. Secondary Outcome: Change From Baseline in Biochemistry - Alkaline Phosphatase (Ratio to Baseline)
Description: Change from baseline (week 0) in alkaline phosphatase (measured in U/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of alkaline phosphatase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 119
Ratio of alkaline phosphatase | 0.94 (15.14) | 0.92 (20.54) | 0.95 (17.83) | 0.95 (13.83)

34. Secondary Outcome: Change From Baseline in Biochemistry - Total Bilirubin (Ratio to Baseline)
Description: Change from baseline (week 0) in total bilirubin (measured in mg/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total bilirubin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 117
Ratio of total bilirubin | 0.89 (34.97) | 0.84 (32.62) | 0.85 (41.55) | 0.95 (39.68)

35. Secondary Outcome: Change From Baseline in Biochemistry - Amylase (Ratio to Baseline)
Description: Change from baseline (week 0) in amylase (measured in U/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 119
Ratio of amylase | 1.09 (23.53) | 1.20 (27.17) | 1.11 (21.64) | 1.05 (26.52)

36. Secondary Outcome: Change From Baseline in Biochemistry - Lipase (Ratio to Baseline)
Description: Change from baseline (week 0) in lipase (measured in U/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 119
Ratio of lipase | 1.24 (43.99) | 1.60 (55.40) | 1.35 (51.48) | 1.05 (32.22)

37. Secondary Outcome: Change From Baseline in Biochemistry - Creatine Kinase (Ratio to Baseline)
Description: Change from baseline (week 0) in creatine kinase (measured in U/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatine kinase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 118
Ratio of creatine kinase | 1.06 (67.51) | 0.96 (48.18) | 1.00 (46.25) | 0.93 (58.87)

38. Secondary Outcome: Change From Baseline in Calcium (Ratio to Baseline)
Description: Change from baseline (week 0) in calcium (measured in mg/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcium
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 119
Ratio of calcium | 0.98 (6.66) | 0.97 (4.87) | 0.98 (4.52) | 0.97 (3.79)

39. Secondary Outcome: Change From Baseline in Potassium (Ratio to Baseline)
Description: Change from baseline (week 0) in potassium (measured in milliequivalents per liter [mEq/L]) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of potassium
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 119 | 121 | 114 | 118
Ratio of potassium | 1.02 (9.73) | 1.01 (8.96) | 1.00 (9.94) | 1.01 (9.98)

40. Secondary Outcome: Change From Baseline in Sodium (Ratio to Baseline)
Description: Change from baseline (week 0) in sodium (measured in mEq/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of sodium
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 119 | 122 | 114 | 118
Ratio of sodium | 1.00 (1.49) | 1.00 (1.46) | 1.00 (1.42) | 1.00 (1.32)

41. Secondary Outcome: Change From Baseline in Albumin (Ratio to Baseline)
Description: Change from baseline (week 0) in albumin (measured in g/dL) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of albumin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 114 | 119
Ratio of albumin | 1.00 (4.07) | 0.99 (4.73) | 0.99 (4.41) | 0.99 (3.95)

42. Secondary Outcome: Change From Baseline in Calcitonin (Ratio to Baseline)
Description: Change from baseline (week 0) in calcitonin (measured in picograms per milliliter [pg/mL]) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 119 | 116 | 118
Ratio of calcitonin | 1.01 (23.53) | 1.09 (39.69) | 1.15 (42.68) | 0.98 (46.93)

43. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from baseline (week 0) in pulse rate at week 26 is presented. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 116 | 121
Beats per minute (beats/min) | 2 (9) | 4 (9) | 5 (9) | 1 (9)

44. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Change from baseline (week 0) in systolic blood pressure at week 26 is presented. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 116 | 121
millimeters of mercury (mmHg) | 1 (13) | -2 (12) | -4 (13) | -2 (13)

45. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Change from baseline (week 0) in diastolic blood pressure at week 26 is presented. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 116 | 121
mmHg | 0 (9) | -1 (8) | -2 (9) | -2 (9)

46. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Category
Description: Change from baseline (week 0) in ECG category at week 26 is presented. Change from baseline results are presented as shift in findings categorized as: normal, abnormal and not clinically significant (NCS), and abnormal and clinically significant (CS). The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, follow-up prematurely discontinuation visit, last dose of trial product plus 38 days or the end-date for the in-trial observation period.
Time Frame: Baseline (Week 0), Week 26
Population: Safety analysis set included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = participants with available data for this outcome measure and Number Analyzed = number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 123 | 119 | 121
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 66 | 75 | 69 | 66
  Normal (week 0) to normal (week 26) | 53 | 61 | 59 | 58
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 66 | 75 | 69 | 66
  Normal (week 0) to abnormal NCS (week 26) | 12 | 11 | 9 | 5
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 66 | 75 | 69 | 66
  Normal (week 0) to abnormal CS (week 26) | 1 | 3 | 1 | 3
  Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 37 | 34 | 43 | 45
  Abnormal NCS (week 0) to normal (week 26) | 9 | 11 | 19 | 12
  Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 37 | 34 | 43 | 45
  Abnormal NCS (week 0) to abnormal NCS (week 26) | 26 | 23 | 23 | 33
  Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 37 | 34 | 43 | 45
  Abnormal NCS (week 0) to abnormal CS (week 26) | 2 | 0 | 1 | 0
  Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 18 | 14 | 7 | 10
  Abnormal CS (week 0) to normal (week 26) | 6 | 4 | 2 | 5
  Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 18 | 14 | 7 | 10
  Abnormal CS (week 0) to abnormal NCS (week 26) | 1 | 1 | 1 | 1
  Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 18 | 14 | 7 | 10
  Abnormal CS (week 0) to abnormal CS (week 26) | 11 | 9 | 4 | 4

47. Secondary Outcome: Change From Baseline in Physical Examination Category
Description: Change from baseline (week 0) in physical examination category at week 26 is presented. The physical examination shift in findings were categorized as normal, abnormal NCS and abnormal CS and are presented for the following body systems: cardiovascular system; central and peripheral nervous system; gastrointestinal system, including mouth; general appearance; head, ears, eyes, nose, throat, neck; lymph node palpation; musculoskeletal system; respiratory system; skin; and thyroid gland. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the last date on trial product plus 3 days.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 121 | 122 | 116 | 121
Participants
  Cardiovascular system - Normal (week 0) to normal (week 26): number analyzed (Participants) | 113 | 118 | 115 | 116
  Cardiovascular system - Normal (week 0) to normal (week 26) | 113 | 118 | 115 | 115
  Cardiovascular system - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 113 | 118 | 115 | 116
  Cardiovascular system - Normal (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 1
  Cardiovascular system - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 113 | 118 | 115 | 116
  Cardiovascular system - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Cardiovascular system - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 8 | 4 | 1 | 4
  Cardiovascular system - Abnormal NCS (week 0) to normal (week 26) | 3 | 2 | 0 | 0
  Cardiovascular system - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 8 | 4 | 1 | 4
  Cardiovascular system - Abnormal NCS (week 0) to abnormal NCS (week 26) | 5 | 2 | 1 | 4
  Cardiovascular system - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 8 | 4 | 1 | 4
  Cardiovascular system - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Cardiovascular system - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 0 | 0 | 1
  Cardiovascular system - Abnormal CS (week 0) to normal (week 26) |  |  |  | 0
  Cardiovascular system - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 1
  Cardiovascular system - Abnormal CS (week 0) to abnormal NCS (week 26) |  |  |  | 0
  Cardiovascular system - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 1
  Cardiovascular system - Abnormal CS (week 0) to abnormal CS (week 26) |  |  |  | 1
  Central and Peripheral Nervous System - Normal (week 0) to normal (week 26): number analyzed (Participants) | 119 | 121 | 116 | 120
  Central and Peripheral Nervous System - Normal (week 0) to normal (week 26) | 119 | 121 | 116 | 120
  Central and Peripheral Nervous System - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 119 | 121 | 116 | 120
  Central and Peripheral Nervous System - Normal (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Central and Peripheral Nervous System - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 119 | 121 | 116 | 120
  Central and Peripheral Nervous System - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Central and Peripheral Nervous System - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 2 | 0 | 0 | 1
  Central and Peripheral Nervous System - Abnormal NCS (week 0) to normal (week 26) | 0 |  |  | 0
  Central and Peripheral Nervous System - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 2 | 0 | 0 | 1
  Central and Peripheral Nervous System - Abnormal NCS (week 0) to abnormal NCS (week 26) | 2 |  |  | 1
  Central and Peripheral Nervous System - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 2 | 0 | 0 | 1
  Central and Peripheral Nervous System - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 |  |  | 0
  Central and Peripheral Nervous System - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 1 | 0 | 0
  Central and Peripheral Nervous System - Abnormal CS (week 0) to normal (week 26) |  | 0 |  |
  Central and Peripheral Nervous System - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 1 | 0 | 0
  Central and Peripheral Nervous System - Abnormal CS (week 0) to abnormal NCS (week 26) |  | 0 |  |
  Central and Peripheral Nervous System - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 1 | 0 | 0
  Central and Peripheral Nervous System - Abnormal CS (week 0) to abnormal CS (week 26) |  | 1 |  |
  Gastrointestinal System incl. Mouth - Normal (week 0) to normal (week 26): number analyzed (Participants) | 118 | 117 | 114 | 115
  Gastrointestinal System incl. Mouth - Normal (week 0) to normal (week 26) | 117 | 117 | 114 | 115
  Gastrointestinal System incl. Mouth - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 118 | 117 | 114 | 115
  Gastrointestinal System incl. Mouth - Normal (week 0) to abnormal NCS (week 26) | 1 | 0 | 0 | 0
  Gastrointestinal System incl. Mouth - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 118 | 117 | 114 | 115
  Gastrointestinal System incl. Mouth - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Gastrointestinal System incl. Mouth - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 3 | 3 | 2 | 5
  Gastrointestinal System incl. Mouth - Abnormal NCS (week 0) to normal (week 26) | 2 | 0 | 0 | 0
  Gastrointestinal System incl. Mouth - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 3 | 3 | 2 | 5
  Gastrointestinal System incl. Mouth - Abnormal NCS (week 0) to abnormal NCS (week 26) | 1 | 3 | 2 | 5
  Gastrointestinal System incl. Mouth - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 3 | 3 | 2 | 5
  Gastrointestinal System incl. Mouth - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Gastrointestinal System incl. Mouth - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 2 | 0 | 1
  Gastrointestinal System incl. Mouth - Abnormal CS (week 0) to normal (week 26) |  | 0 |  | 0
  Gastrointestinal System incl. Mouth - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0. | 2 | 0 | 1
  Gastrointestinal System incl. Mouth - Abnormal CS (week 0) to abnormal NCS (week 26) |  | 0 |  | 0
  Gastrointestinal System incl. Mouth - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 2 | 0 | 1
  Gastrointestinal System incl. Mouth - Abnormal CS (week 0) to abnormal CS (week 26) |  | 2 |  | 1
  General Appearance - Normal (week 0) to normal (week 26): number analyzed (Participants) | 116 | 118 | 110 | 119
  General Appearance - Normal (week 0) to normal (week 26) | 115 | 118 | 110 | 119
  General Appearance - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 116 | 118 | 110 | 119
  General Appearance - Normal (week 0) to abnormal NCS (week 26) | 1 | 0 | 0 | 0
  General Appearance - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 116 | 118 | 110 | 119
  General Appearance - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  General Appearance - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 4 | 4 | 5 | 1
  General Appearance - Abnormal NCS (week 0) to normal (week 26) | 4 | 2 | 1 | 0
  General Appearance - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 4 | 4 | 5 | 1
  General Appearance - Abnormal NCS (week 0) to abnormal NCS (week 26) | 0 | 2 | 4 | 1
  General Appearance - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 4 | 4 | 5 | 1
  General Appearance - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  General Appearance - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 1 | 0 | 1 | 1
  General Appearance - Abnormal CS (week 0) to normal (week 26) | 0 |  | 0 | 0
  General Appearance - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 1 | 0 | 1 | 1
  General Appearance - Abnormal CS (week 0) to abnormal NCS (week 26) | 0 |  | 0 | 0
  General Appearance - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 1 | 0 | 1 | 1
  General Appearance - Abnormal CS (week 0) to abnormal CS (week 26) | 1 |  | 1 | 1
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (week 0) to normal (week 26): number analyzed (Participants) | 121 | 118 | 115 | 118
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (week 0) to normal (week 26) | 121 | 118 | 115 | 117
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 121 | 118 | 115 | 118
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 121 | 118 | 115 | 118
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 1
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 1 | 0 | 2
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (week 0) to normal (week 26) |  | 0 |  | 1
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 1 | 0 | 2
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (week 0) to abnormal NCS (week 26) |  | 1 |  | 1
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 1 | 0 | 2
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (week 0) to abnormal CS (week 26) |  | 0 |  | 0
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 3 | 1 | 1
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (week 0) to normal (week 26) |  | 0 | 0 | 0
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 3 | 1 | 1
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (week 0) to abnormal NCS (week 26) |  | 0 | 0 | 0
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 3 | 1 | 1
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (week 0) to abnormal CS (week 26) |  | 3 | 1 | 1
  Lymph Node Palpation - Normal (week 0) to normal (week 26): number analyzed (Participants) | 120 | 121 | 115 | 119
  Lymph Node Palpation - Normal (week 0) to normal (week 26) | 120 | 121 | 115 | 119
  Lymph Node Palpation - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 120 | 121 | 115 | 119
  Lymph Node Palpation - Normal (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Lymph Node Palpation - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 120 | 121 | 115 | 119
  Lymph Node Palpation - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Lymph Node Palpation - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 1 | 1 | 1 | 2
  Lymph Node Palpation - Abnormal NCS (week 0) to normal (week 26) | 1 | 1 | 1 | 2
  Lymph Node Palpation - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 1 | 1 | 1 | 2
  Lymph Node Palpation - Abnormal NCS (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Lymph Node Palpation - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 1 | 1 | 1 | 2
  Lymph Node Palpation - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Lymph Node Palpation - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Lymph Node Palpation - Abnormal CS (week 0) to abnormal NCS (week 26)0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lymph Node Palpation - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Musculoskeletal System - Normal (week 0) to normal (week 26): number analyzed (Participants) | 120 | 119 | 115 | 120
  Musculoskeletal System - Normal (week 0) to normal (week 26) | 119 | 119 | 115 | 119
  Musculoskeletal System - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 120 | 119 | 115 | 120
  Musculoskeletal System - Normal (week 0) to abnormal NCS (week 26) | 1 | 0 | 0 | 0
  Musculoskeletal System - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 120 | 119 | 115 | 120
  Musculoskeletal System - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 1
  Musculoskeletal System - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 1 | 1 | 1 | 0
  Musculoskeletal System - Abnormal NCS (week 0) to normal (week 26) | 0 | 0 | 0 |
  Musculoskeletal System - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 1 | 1 | 1 | 0
  Musculoskeletal System - Abnormal NCS (week 0) to abnormal NCS (week 26) | 1 | 1 | 1 |
  Musculoskeletal System - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 1 | 1 | 1 | 0
  Musculoskeletal System - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 |
  Musculoskeletal System - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 2 | 0 | 1
  Musculoskeletal System - Abnormal CS (week 0) to normal (week 26) |  | 1 |  | 0
  Musculoskeletal System - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 2 | 0 | 1
  Musculoskeletal System - Abnormal CS (week 0) to abnormal NCS (week 26) |  | 0 |  | 0
  Musculoskeletal System - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 2 | 0 | 1
  Musculoskeletal System - Abnormal CS (week 0) to abnormal CS (week 26) |  | 1 |  | 1
  Respiratory System - Normal (week 0) to normal (week 26) | 121 | 122 | 116 | 121
  Respiratory System - Normal (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Respiratory System - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Respiratory System - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Respiratory System - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Respiratory System - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Respiratory System - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Respiratory System - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Respiratory System - Abnormal CS (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Respiratory System - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 0
  Skin - Normal (week 0) to normal (week 26): number analyzed (Participants) | 101 | 106 | 99 | 105
  Skin - Normal (week 0) to normal (week 26) | 99 | 106 | 98 | 105
  Skin - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 101 | 106 | 99 | 105
  Skin - Normal (week 0) to abnormal NCS (week 26) | 1 | 0 | 1 | 0
  Skin - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 101 | 106 | 99 | 105
  Skin - Normal (week 0) to abnormal CS (week 26) | 1 | 0 | 0 | 0
  Skin - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 13 | 7 | 14 | 12
  Skin - Abnormal NCS (week 0) to normal (week 26) | 2 | 0 | 3 | 3
  Skin - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 13 | 7 | 14 | 12
  Skin - Abnormal NCS (week 0) to abnormal NCS (week 26) | 11 | 7 | 11 | 9
  Skin - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 13 | 7 | 14 | 12
  Skin - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Skin - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 7 | 9 | 3 | 4
  Skin - Abnormal CS (week 0) to normal (week 26) | 0 | 2 | 1 | 1
  Skin - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 7 | 9 | 3 | 4
  Skin - Abnormal CS (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Skin - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 7 | 9 | 3 | 4
  Skin - Abnormal CS (week 0) to abnormal CS (week 26) | 7 | 7 | 2 | 3
  Thyroid Gland - Normal (week 0) to normal (week 26): number analyzed (Participants) | 119 | 120 | 113 | 119
  Thyroid Gland - Normal (week 0) to normal (week 26) | 119 | 120 | 113 | 119
  Thyroid Gland - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 119 | 120 | 113 | 119
  Thyroid Gland - Normal (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Thyroid Gland - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 119 | 120 | 113 | 119
  Thyroid Gland - Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Thyroid Gland - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 2 | 2 | 3 | 1
  Thyroid Gland - Abnormal NCS (week 0) to normal (week 26) | 0 | 0 | 0 | 0
  Thyroid Gland - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 2 | 2 | 3 | 1
  Thyroid Gland - Abnormal NCS (week 0) to abnormal NCS (week 26) | 2 | 2 | 3 | 1
  Thyroid Gland - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 2 | 2 | 3 | 1
  Thyroid Gland - Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0
  Thyroid Gland - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 0 | 0 | 0 | 1
  Thyroid Gland - Abnormal CS (week 0) to normal (week 26) |  |  |  | 0
  Thyroid Gland - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 1
  Thyroid Gland - Abnormal CS (week 0) to abnormal NCS (week 26) |  |  |  | 0
  Thyroid Gland - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 0 | 0 | 0 | 1
  Thyroid Gland - Abnormal CS (week 0) to abnormal CS (week 26) |  |  |  | 1

48. Secondary Outcome: Change From Baseline in Eye Examination Category
Description: Change from baseline (week 0) in eye examination category at week 26 is presented. Eye examination shift in findings were categorized as normal, abnormal NCS and abnormal CS. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, follow-up prematurely discontinuation visit, last date on trial product plus 38 days or the end-date for the in-trial observation period.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 120 | 121 | 119 | 121
Participants
  Left Eye Ophthalmoscopy - Normal (week 0) to normal (week 26): number analyzed (Participants) | 81 | 86 | 90 | 85
  Left Eye Ophthalmoscopy - Normal (week 0) to normal (week 26) | 73 | 77 | 83 | 75
  Left Eye Ophthalmoscopy - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 81 | 86 | 90 | 85
  Left Eye Ophthalmoscopy - Normal (week 0) to abnormal NCS (week 26) | 6 | 5 | 5 | 5
  Left Eye Ophthalmoscopy - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 81 | 86 | 90 | 85
  Left Eye Ophthalmoscopy - Normal (week 0) to abnormal CS (week 26) | 2 | 4 | 2 | 5
  Left Eye Ophthalmoscopy - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 29 | 23 | 17 | 20
  Left Eye Ophthalmoscopy - Abnormal NCS (week 0) to normal (week 26) | 10 | 2 | 1 | 2
  Left Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 29 | 23 | 17 | 20
  Left Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal NCS (week 26) | 15 | 19 | 15 | 18
  Left Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 29 | 23 | 17 | 20
  Left Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal CS (week 26) | 4 | 2 | 1 | 0
  Left Eye Ophthalmoscopy - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 10 | 12 | 12 | 16
  Left Eye Ophthalmoscopy - Abnormal CS (week 0) to normal (week 26) | 2 | 4 | 4 | 7
  Left Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 10 | 12 | 12 | 16
  Left Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal NCS (week 26) | 0 | 1 | 0 | 0
  Left Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 10 | 12 | 12 | 16
  Left Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal CS (week 26) | 8 | 7 | 8 | 9
  Right Eye Ophthalmoscopy - Normal (week 0) to normal (week 26): number analyzed (Participants) | 85 | 86 | 89 | 82
  Right Eye Ophthalmoscopy - Normal (week 0) to normal (week 26) | 76 | 76 | 82 | 74
  Right Eye Ophthalmoscopy - Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 85 | 86 | 89 | 82
  Right Eye Ophthalmoscopy - Normal (week 0) to abnormal NCS (week 26) | 6 | 6 | 4 | 5
  Right Eye Ophthalmoscopy - Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 85 | 86 | 89 | 82
  Right Eye Ophthalmoscopy - Normal (week 0) to abnormal CS (week 26) | 3 | 4 | 3 | 3
  Right Eye Ophthalmoscopy - Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 26 | 22 | 19 | 22
  Right Eye Ophthalmoscopy - Abnormal NCS (week 0) to normal (week 26) | 8 | 3 | 3 | 3
  Right Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 26 | 22 | 19 | 22
  Right Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal NCS (week 26) | 14 | 18 | 15 | 19
  Right Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 26 | 22 | 19 | 22
  Right Eye Ophthalmoscopy - Abnormal NCS (week 0) to abnormal CS (week 26) | 4 | 1 | 1 | 0
  Right Eye Ophthalmoscopy - Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 9 | 13 | 11 | 17
  Right Eye Ophthalmoscopy - Abnormal CS (week 0) to normal (week 26) | 2 | 3 | 5 | 8
  Right Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 9 | 13 | 11 | 17
  Right Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal NCS (week 26) | 0 | 1 | 1 | 0
  Right Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 9 | 13 | 11 | 17
  Right Eye Ophthalmoscopy - Abnormal CS (week 0) to abnormal CS (week 26) | 7 | 9 | 5 | 9

49. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. TEAE was defined as an AE with onset in the on-treatment observation period. On-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, follow-up prematurely discontinuation visit, last date on trial product plus 38 days or the end-date for the in-trial observation period.
Time Frame: Up to 31 weeks
Population: Safety analysis set included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 129 | 131
Events | 251 | 292 | 231 | 212

50. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemia was defined as an episode that was severe according to the ADA classification or BG confirmed by a plasma glucose (PG) value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, follow-up prematurely discontinuation visit, last date on trial product plus 38 days or the end-date for the in-trial observation period.
Time Frame: Up to 31 weeks
Population: Safety analysis set included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 129 | 131
Episodes | 0 | 0 | 0 | 0

51. Secondary Outcome: Number of Participants With Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: as for outcome 50
Time Frame: Up to 31 weeks
Population: Safety analysis set included all participants exposed to at least one dose of trial product.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 129 | 131
Participants | 0 | 0 | 0 | 0

52. Secondary Outcome: Anti-semaglutide Binding Antibody Levels
Description: Anti-semaglutide binding antibody levels measured anytime during post-baseline visits (week 0 to week 31) are presented. The outcome data are presented as percentage of bound radioactivity-labelled semaglutide/total added radioactivity-labelled semaglutide (%B/T). Results are based on the data from the in-trial observation period - the in-trial observation period started at randomization and ended at the date of: the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact, and death for participants who died before any of the above.
Time Frame: Up to 31 weeks
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 0 | 1 | 0
%B/T |  | 2.1 |

53. Secondary Outcome: Number of Participants With Anti-semaglutide Binding Antibodies
Description: Number of participants who had anti-semaglutide binding antibody levels anytime during post-baseline visits (week 0 to week 31) are presented. Results are based on the data from the in-trial observation period - the in-trial observation period started at randomization and ended at the date of: the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participants-investigator contact, and death for participants who died before any of the above.
Time Frame: Up to 31 weeks
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 91 | 93 | 85
Participants | 0 | 1 | 0

54. Secondary Outcome: Number of Participants With Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1
Description: Number of participants who had anti-semaglutide binding antibodies cross reacting with native glucagon-like peptide-1 (GLP-1) anytime during post-baseline visits (week 0 to week 31) are presented. Results are based on the data from the in-trial observation period - the in-trial observation period started at randomization and ended at the date of: the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact, and death for participants who died before any of the above.
Time Frame: Up to 31 weeks
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 91 | 93 | 85
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From week 0 to week 31
Description: All presented adverse events (AEs) are treatment-emergent (i.e., TEAEs). TEAE was defined as an AE with onset in the on-treatment observation period.
  Results are based on the safety analysis set (SAS) which included all participants exposed to at least one dose of trial product.
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/130 | 0/129 | 0/131
Serious Adverse Events (participants affected / at risk) | 6/130 | 10/130 | 5/129 | 2/131
Other Adverse Events (participants affected / at risk) | 30/130 | 47/130 | 40/129 | 16/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=130) | Oral Semaglutide 7 mg (N=130) | Oral Semaglutide 14 mg (N=129) | Placebo (N=131)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=130) | Oral Semaglutide 7 mg (N=130) | Oral Semaglutide 14 mg (N=129) | Placebo (N=131)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 10 (13) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 6 (7) | 14 (14) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 12 (16) | 12 (18) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 7 (7)
Lipase increased (Investigations) | 7 (12) | 11 (12) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 8 (8) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 12 (14) | 9 (12) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04109547/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT04109547/SAP_001.pdf